CLINICAL TRIAL: NCT05034848
Title: Peripheral Artery Disease (PAD) : Its Effects on Bone
Acronym: AMICOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no practitionner
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2018-13
Record Dates: First submitted 2020-02-19; First posted 2021-09-05 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Bone; Peripheral Artery Disease
Keywords: bone; osteoporosis; peripheral artery disease; HRpQCT
MeSH Terms: conditions — Peripheral Arterial Disease; Osteoporosis

STUDY DESIGN:
Intervention Model Description: observational, interventional, non comparative, prospective, monocentric open study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAD group (Other): PAD patients, diagnosis after undergoing an echo-doppler in the Vascular Medicine Department of Orleans regional Hospital
  Interventions: Procedure: Assessment of BMD by DXA and HRpQCT

INTERVENTIONS:
Procedure: Assessment of BMD by DXA and HRpQCT — * DXA : BMD assessment at the left hip, rachis and both legs
  * HRpQCT : Volumic Bone mineral density, cortical and trabecular parameters, at the non dominant radius and legs
  * Biological samples

SUMMARY:
Prevalence of PAD and osteoporosis (OP) both get higher with age. Clinical and epidemiologic evidence have showed an increased cardiovascular risk in OP and bone loss and fragility fractures in patient with cardiovascular disease.

This study will examine the relationship between vascular disease in legs and sBMD and vBMD at trabecular and cortical sites and bone microarchitecture.

DETAILED DESCRIPTION:
The primary goal of our study is to determinate if presence of PAD is associated with lower sBMD and vBMD values at the tibias, assuming that BMD should be more alterate in the predominant vascular impairement site.

Our secondary objectives are to :

* determine if severity of PAD quantified by ankle brachial index ABI is associated to a decrease of BMD values defined by T-Score at the left hip, spine and legs, but also with volumetric values, assessed by HRpQCT at the non dominant radius and at both tibias.
* determine the prevalence of osteoporosis in our population
* To evaluate the relationships between ;
* lipids and bone parameters
* vit D and parathormone with PAD severity
* levels of physical activity and both vascular and bone impairments

ELIGIBILITY:
Inclusion Criteria:

* PAD patients defined by an Ankle brachial index < 0.9
* Written consent
* Patient affiliated with a social security organism

Exclusion Criteria:

* Age < 18 years
* Pregnancy or risk of pregnancy
* Patients Under guardianship
* Patient with known PAD who had been previously treated by surgery or endovascular pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) volumic values at the tibias of PAD (Peripheral Artery Disease) patients | Day 0
  BMD volumic values are BMD volumetric bone mineral density (mg HA/cm3)

SECONDARY OUTCOMES:
Bone Mineral Density (BMD) measurement by DXA | Day 0
  Relations between areal BMD results (DXA) at the hip and lumbar spine and the ankle brachial index measured at the two legs.
Correlation between microstructural parameters and ankle brachial index results | Day 0
  The following micro structural parameters assessed by HRpQCT at both tibias will be :
  * Dtrab : volumetric trabecular bone mineral density (mg HA/ cm3),
  * Dinn : inner trabecular bone density (mg HA/cm3),
  * Dmeta: metatrabecular bone density (mg HA/cm3),
  * Dcort: volumetric cortical bone mineral density (mg HA/cm3),
  * D100: total volumetric bone mineral density (mg HA/cm3),
  * Tb.Th: trabecular thickness (mm),
  * Tb.N: trabecular number (mm-1);
  * Tb.Sp: trabecular separation (mm),
  * Ct.Th: cortical thickness (mm);
  * Tb1.NSD: intra-distribution individual separation (mm),
  * BV / TV: trabecular bone volume (%).
Comparison between microstructural parameters at tibias | Day 0
  comparison between bone microarchitecture parameters at the tibia: the parameters will be compared between the most severely limb and the contralateral one.
Correlation between Lipid and bone parameters | Day 0
  We will study the relation between lipidic and bone parameters. Potential correlations between on the one hand (lipid parameters: total and HDL-cholesterol, triglyceridemia, LDL-cholesterol calculation) and on the other hand bone parameters: vBMD volumetric bone mineral density (mg HA/cm3) Ct.BMD: cortical volumetric bone mineral density (mg/cm3); Tb.BMD: trabecular volumetric bone mineral density (mg HA/cm3)
Percentage of densitometric osteoporotic patients | Day 0
  percentage of densitometric osteoporotic patients in the population
Evaluation of risk of fracture | Day 0
  The risk of fracture at 10 years will be evaluate by the Fracture Risk Assessment Tool (FRAX) survey.
  The FRAX® tool was developed by the then WHO Collaborating Centre for Metabolic Bone Diseases (1991-2010) at the University of Sheffield. It was launched in 2008 following approximately 10 years of meta-analyses of a variety of risk factors for osteoporotic fracture. Although not the only fracture prediction tool available, FRAX® is the only risk calculator which has been calibrated to rates of fracture and mortality per individual country and has been shown to identify a risk amenable to available treatments.
Evaluation of cardiovascular risk | Day 0
  Cardiovascular risk assessment using the SCORE tool (Systematic Coronary Risk Estimation).
  Four levels of risk are defined:
  * Very high cardiovascular risk ≥ 10%;
  * High risk, which includes subjects with major or particularly high risk factors (familial hypercholesterolemia, severe hypertension, etc.) and those with a score between 5 and 10%;
  * Moderate risk, which concerns patients with a score between 1 and 5%;
  * Low risk, which includes subjects with a score < 1%;
Correlation between microstructural parameters at tibias and radius | Day 0
  comparison between bone microarchitecture at the tibia and of the radius.
  The following micro structural parameters assessed by HRpQCT at tibias and radius will be :
  * Dtrab : volumetric trabecular bone mineral density (mg HA/ cm3),
  * Dinn : inner trabecular bone density (mg HA/cm3),
  * Dmeta: metatrabecular bone density (mg HA/cm3),
  * Dcort: volumetric cortical bone mineral density (mg HA/cm3),
  * D100: total volumetric bone mineral density (mg HA/cm3),
  * Tb.Th: trabecular thickness (mm),
  * Tb.N: trabecular number (mm-1);
  * Tb.Sp: trabecular separation (mm),
  * Ct.Th: cortical thickness (mm);
  * Tb1.NSD: intra-distribution individual separation (mm),
  * BV / TV: trabecular bone volume (%).

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSAILLES, Dr, Principal Investigator — CHR Orleans
Locations (1):
- CHR d'ORLEANS, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breban S, Benhamou CL, Chappard C. Dual-energy X-ray absorptiometry assessment of tibial mid-third bone mineral density in young athletes. J Clin Densitom. 2009 Jan-Mar;12(1):22-7. doi: 10.1016/j.jocd.2008.10.009. Epub 2008 Dec 25. PMID 19111489
- [Background] Collins TC, Ewing SK, Diem SJ, Taylor BC, Orwoll ES, Cummings SR, Strotmeyer ES, Ensrud KE; Osteoporotic Fractures in Men (MrOS) Study Group. Peripheral arterial disease is associated with higher rates of hip bone loss and increased fracture risk in older men. Circulation. 2009 May 5;119(17):2305-12. doi: 10.1161/CIRCULATIONAHA.108.820993. Epub 2009 Apr 20. PMID 19380619
- [Background] Fehervari M, Sarkadi H, Krepuska M, Sotonyi P, Acsady G, Entz L, Lakatos P, Szeberin Z. Bone mineral density is associated with site-specific atherosclerosis in patients with severe peripheral artery disease. Calcif Tissue Int. 2013 Jul;93(1):55-61. doi: 10.1007/s00223-013-9727-5. Epub 2013 Apr 6. PMID 23564349
- [Background] Gaudio A, Muratore F, Fiore V, Rapisarda R, Signorelli SS, Fiore CE. Decreased bone cortical density at the forearm in subjects with subclinical peripheral arterial disease. Osteoporos Int. 2015 Jun;26(6):1747-53. doi: 10.1007/s00198-015-3057-6. Epub 2015 Feb 12. PMID 25672808